CLINICAL TRIAL: NCT02599168
Title: The Effect of Dexmedetomidine on Propofol Requirements During Anesthesia Administered by Bispectral Index-Guided Closed-Loop Anesthesia Delivery System: A Randomized Controlled Study
Brief Title: Effect of Dexmedetomidine on Propofol Requirement During Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr Nitin Sethi (Other)
Responsible Party: Sponsor-Investigator, Dr Nitin Sethi, Doctor, Sir Ganga Ram Hospital
Organization: Sir Ganga Ram Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: EC/04/15/807
Record Dates: First submitted 2015-10-28; First posted 2015-11-06 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Anesthesia
Keywords: dexmedetomidine; propofol; BIS; CLADS
MeSH Terms: interventions — Propofol; Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine group (Active Comparator): Patients will receive a pre-induction loading dose of dexmedetomidine 1-µ/kg over 10 minutes followed by an intraoperative infusion of 0.5-µ/kg/hour . Over and above the use of study drug dexmedetomidine propofol administration will be controlled with Closed Loop Anaesthesia Delivery system to maintain a consistent anaesthetic depth (BIS 40-60) using bispectral index monitor in all the patients
  Interventions: Drug: Propofol; Drug: Dexmedetomidine
- Non-Dexmedetomidine group (Placebo Comparator): Patients will receive a pre-induction loading dose of 0.9% saline solution over 10 minutes followed by an intraoperative infusion.Over and above the use of 0.9% saline solution propofol administration will be controlled with Closed Loop Anaesthesia Delivery system to maintain a consistent anaesthetic depth (BIS 40-60) using bispectral index monitor in all the patients
  Interventions: Drug: Propofol; Drug: Placebo (normal saline)

INTERVENTIONS:
Drug: Propofol
Drug: Dexmedetomidine
  Arms: Dexmedetomidine group
Drug: Placebo (normal saline)
  Arms: Non-Dexmedetomidine group

SUMMARY:
Dexmedetomidine, a selective alpha-2 agonist agent used for maintaining sedation in intensive care patients in receipt of mechanical ventilation, is being increasingly utilized in anaesthesia practice for facilitating anaesthesia depth as an adjunct to base anaesthetics (intravenous; propofol: inhalational; sevoflurane, desflurane). The investigators intend to assess the anaesthetic potential of dexmedetomidine in controlled anaesthesia settings empowered by the use of an objective, patient response based, safe, efficient, and patented closed loop anaesthesia delivery system (CLADS). CLADS functions on control of processed EEG response parameter captured from anaesthetized patients with the help of a BIS- monitor, which is continuously fed into a automated drug infusion pump. The infusion pump then accordingly delivers the anaesthetic drug to the patients based on pharmacodynamic requirements. If dexmedetomidine has anaesthesia potential then it is likely that propofol use delivered by CLADS can be reduced further. In addition the effect of two drugs (viz, base agent-propofol plus adjunct agent-dexmedetomidine) on different receptor site within the brain would help gain greater anaesthetic depth consistency as well as a lower incidence of intraoperative patient awareness. This prospective randomized two-arm study aims to assess effect of the use of dexmedetomidine on propofol requirements (primary objective), anaesthesia depth consistency, and intraoperative patient awareness (secondary objectives).

DETAILED DESCRIPTION:
After Institutional Ethics Committee approval and written informed consent, eighty patient-participants (40 per group) aged 20-65 years, ASA physical status I/II, of either sex, and undergoing major laparoscopic / robotic surgery of more than 60-minutes duration will be included in this single-center (Sir Ganga Ram Hospital, New Delhi-110060, India ) prospective, double-blinded, two-arm, randomized controlled study.

The patients will be randomly divided into two groups:

Group-I: Pre-induction dexmedetomidine + intraoperative dexmedetomidine plus anesthesia with propofol delivered by CLADS (induction + maintenance) [Dexmedetomidine group] Group-II: Pre-induction 0.9% saline solution + intraoperative 0.9% saline solution infusion + anesthesia with propofol delivered by CLADS (induction + maintenance) [Non Dexmedetomidine group]

Sample-size Estimation:

The sample size estimation was estimated from the cue that the average propofol doses required for maintenance of anaesthesia (4.7+ 1.6 mg/kg/hr) when using manual propofol and remifentanil target controlled infusion18 with a 90% power employed to detect a 30% decrease of propofol dosage among the patients who will receive dexmedetomidine in addition to base anesthetic propofol; with a bilateral α risk value of 0.05, the investigators would require 66 patients for the study. To cover up for unanticipated losses the investigators would need additional 20% patients. Thus the investigators would require 80-patients for the study

Randomization, Allocation Concealment:

The patients will be randomly allocated to one of the two groups based on a computer-generated random number table (url:stattrek.com/statistics/random-number-generator.aspx). Randomization sequence concealment will include opaque-sealed envelopes with alphabetic codes whose distribution will be in control of an independent analyst. The envelopes will be opened; patient's data-slip will be pasted on them, and will be sent back to the control analyst.

Management of Anaesthesia:

Two peripheral venous lines (18G/20G catheter) will be secured. Invasive vascular access (arterial line for direct continuous blood pressure assessment, central venous catheter) will be secured as per the requirement of surgery and/or patients morbid status. A BIS sensor (Covidien IIc, Mansfield, USA) for monitoring depth of anaesthesia, using the BIS monitoring module (Model DSC-XP, Aspect medical system, USA), will be applied over the patient's forehead according to manufacturer's instruction prior to induction of anaesthesia.

The patients will be randomly allocated to one of the two groups separated by method of dexmedetomidine administration. The pre-induction and the infusion dose of dexmedetomidine will be 1-µ/kg over 10 minutes and 0.5-µ/kg/hour, respectively. Dexmedetomidine infusion will be stopped in case of acute haemodynamic suppression (>20% pre-induction baseline) or acute blood loss (>200-ml) at any point of time and it will be recorded as an event. It will be restarted upon normalcy of haemodynamics is achieved and also full surgical hemostasis is ensured.

Anesthesia Technique:

All the patients will be administered pre-induction fentanyl-citrate analgesia as per a predefined strategy (total 2-µg/kg IV: 1-µg/kg at 0 minute, 3-minutes time points]. Pre-oxygenation will be initiated at 6-minute time point or prior to that if there is a fall in oxygen saturation < 94 percent. At 9-minute time point anaesthesia will be induced with propofol 2-mg/kg and vecuronium bromide 0.08-mg/kg for skeletal muscle relaxation to facilitate tracheal intubation. Ventilator settings of CMV, tracheal tube size [7.5-mm I.D (male), 6.5-mm I.D (female)] and breathing circuit (circle-CO2 absorber system) will be the standardized in all the patients. Routine monitoring (EKG, NIBP, pulse oximetery, EtCO2) will be applied during the procedure as per the established practice. Over and above the use of study drug dexmedetomidine as per group allocation, propofol administration will be controlled with CLADS system tuned to consistent anaesthetic depth (BIS 40-60) in all the patients. In addition, all the patients will receive 0.5-µg/kg/hr fentanyl infusion during surgery. Oxygen.-air mixture (FiO2 0.50) will be utilized for intraoperative ventilation. Neostigmine (50-µg/kg) and glycopyrrolate (20-µg/kg) will be administered to reverse the residual neuromuscular blockade (non-depolariser).

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status I/II
2. Undergoing elective laparoscopic / robotic surgery of more than 60-minutes duration

Exclusion Criteria:

1. Cardiovascular disorders (uncontrolled hypertension, Atrio-ventricular block, sinus bradycardia, congenital heart disease, reduced LV compliance & diastolic dysfunction)
2. Neurological disorders (previous neurosurgery, psychiatric disorders, autonomic nervous system disorders- orthostatic hypotension, transient ischemic attacks)
3. Any hepato-renal insufficiency
4. Uncontrolled diabetes mellitus
5. Known allergy/hypersensitivity to study drug
6. Pulmonary dysfunction (restrictive /obstructive lung disease)
7. Acute/chronic drug dependence/substance abuse

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-12-05 (Actual); Primary Completion 2017-03-20 (Actual); Study Completion 2017-03-20 (Actual)

PRIMARY OUTCOMES:
Change in Propofol usage in milligrams | From beginning of anaesthesia (0-hours, baseline) till 6 hours intraoperatively
  Comparison of 'dexmedetomidine' versus 'no dexmedetomidine' administration in decreasing quantitative propofol requirements (measured in milligrams) during closed loop anaesthesia delivery system empowered and Bi-spectral index controlled propofol-based general anaesthesia.
Assessment of change in anaesthesia depth using Bi-spectral index score | From beginning of anaesthesia (0-hours, baseline) till 6 hours intraoperatively
  Comparison of anaesthesia depth adequacy in intervention (with dexmedetomidine) versus control (without dexmedetomidine) using Varvel criteria to assess Bi-spectral index (BIS) score consistency during closed loop anaesthesia delivery system empowered and BIS-controlled propofol-based general anaesthesia

SECONDARY OUTCOMES:
Change in Intraoperative heart Rate (beats per minute) | From beginning of anaesthesia (0-hours, baseline) till 6 hours intraoperatively
  Comparison of intraoperative heart rate in the 'intervention' (with dexmedetomidine) versus 'control' (without dexmedetomidine) during closed loop anaesthesia delivery system empowered and Bi-spectral index controlled propofol-based GA
Change in Intraoperative blood pressure - systolic , diastolic, and mean (mmHg) | From beginning of anaesthesia (0-hours, baseline) till 6 hours intraoperatively
  Comparison of intraoperative blood pressure (systolic , diastolic, and mean) in the 'intervention' (with dexmedetomidine) versus 'control' (without dexmedetomidine) during closed loop anaesthesia delivery system empowered and Bi-spectral index controlled propofol-based GA
Postoperative sedation | From the end of anaesthesia till 24-hours, postoperatively
  Will be assessed using Observer asssesment of Alertness/Sedation Scale (OAAS)
Intraoperative awareness | From the end of anaesthesia till 48-hours, postoperatively
  Will be assessed using modified brice questionnaire
Postoperative nausea and vomiting | From the end of anaesthesia till 24-hours, postoperatively
  Will be assessed using PONV scale
Postoperative Analgeisa | From the end of anaesthesia till 24-hours, postoperatively
  Will be assessed using Visual Analogue Scale (VAS) Score

CONTACTS AND LOCATIONS:
Overall Officials: Goverdhan D Puri, MD, PhD, Study Director — Post Graduate Institute of Medical Education & Research, Chandigarh, India; Jayashree Sood, MD, FFRCA, Study Chair — Sir Ganga Ram Hospital, New Delhi, INDIA; Amitabh Dutta, MD, Principal Investigator — Sir Ganga Ram Hospital, New Delhi, INDIA
Locations (1):
- Sir Ganga Ram Hospital, New Delhi, India

REFERENCES:
- [Derived] Dutta A, Sethi N, Sood J, Panday BC, Gupta M, Choudhary P, Puri GD. The Effect of Dexmedetomidine on Propofol Requirements During Anesthesia Administered by Bispectral Index-Guided Closed-Loop Anesthesia Delivery System: A Randomized Controlled Study. Anesth Analg. 2019 Jul;129(1):84-91. doi: 10.1213/ANE.0000000000003470. PMID 29787410